CLINICAL TRIAL: NCT04417101
Title: A Prospective Randomized Crossover Trial to Explore the Tolerability, Safety and Effectiveness of Chinese Herbal Medicine Among Patients With Dialysis-related Myofascial Pain
Brief Title: Chinese Herbal Medicine for Dialysis-related Myofascial Pain: Study Protocol for A Pilot Randomized Study
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 202000477A3
Record Dates: First submitted 2020-05-27; First posted 2020-06-04 (Actual); Last update posted 2020-06-04 (Actual); Status verified 2020-05

CONDITIONS: Myofascial Pain Syndrome
MeSH Terms: conditions — Myofascial Pain Syndromes | interventions — Ephedrae herba

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- JBT treatment (Experimental): The participants will be instructed to take their Chinese herbal medicine formula (CHM), which named Juan Bi Tang, and take it as a dose of 3 g (per bag) each time, trice daily for 4 weeks.
  Interventions: Drug: Chinese Herb
- No treatment (No Intervention): Participants in the non-treatment period will receive conventional self-care management for myofascial pain syndrome.

INTERVENTIONS:
Drug: Chinese Herb — The participants will be instructed to take their JBT and take it as a dose of 3 g (per bag) each time, trice daily for 4 weeks.
  Arms: JBT treatment

SUMMARY:
Dialysis-related myofascial pain in hemodialysis (HD) patients is an important issue that is associated with many other psychosomatic problems. Effective interventions are required to alleviate pain problems in this group. Chinese herbal medicine (CHM) has been tried as a potential therapeutic method to improve pain. The aim of this study is to evaluate the effect of a CHM formula intervention on pain intensity, daily function, and quality of life, and safety among HD patients in dialysis center within a southern Taiwan context.

ELIGIBILITY:
Inclusion Criteria:

* Adults (aged ≥ 20 y) undergoing conventional HD three times a week via an AV fistula;
* To have myofascial trigger points (MTrPs) in one or more of the following muscles around the AV fistula: the flexor carpi radialis, palmaris longus, the pronator teres, the palmaris longus, and/or the finger flexor, diagnosed by dialysis-related myofascial pain, which must be experiencing pain during HD [M1];
* Onset of symptoms within 1 month before enrollment;
* Capable of giving adequate response to pain;
* Have an exquisite tenderness was found on palpation in the taut band with moderate intensity of pain at baseline (ie, a pain score > 3 on a numeric rating scale);
* Can commit to not change their medication and dialytic method during the 10 weeks of this study.

Exclusion Criteria:

* Severe chronic or acute disease interfering with attendance for therapy;
* Have comorbid conditions such as rheumatoid arthritis, stroke, tumor, coagulopathy, chronic liver disease, radiculopathies of the upper limb, recent history of cervical/shoulder/arm surgery, or trauma;
* Have depression and/or presence of a psychiatric disorder;
* Have taken painkillers, muscle relaxant, and anti-inflammatory medications or used topical anesthetics in the past week;
* Have allergy to Chinese herbal product;
* Unable to understand or sign an informed consent form.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-07-01 (Estimated); Primary Completion 2021-06-30 (Estimated); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
Quality of life during dialysis | 1 year
  Kidney Disease Quality of Life 36-Item Short-Form Survey

SECONDARY OUTCOMES:
Motor function of upper limb | 1 year
  Fugl-Meyer Assessment for upper extremity
Muscle power | 1 year
  Gripping algometer
Pain score during dialysis | 1 year
  Visual Analogue Scale (0-100)

CONTACTS AND LOCATIONS:
Overall Officials: Ming-Yen C Tsai, Principal Investigator — 長庚紀念醫院

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hsu YT, Ng HY, Chen YH, Huang YC, Lee YY, Tsai MY. Assessing the efficacy and safety of Juan Bi Tang for dialysis-related myofascial pain in the fistula arm: Study protocol for a randomized cross-over trial. Front Public Health. 2022 Aug 19;10:925232. doi: 10.3389/fpubh.2022.925232. eCollection 2022. PMID 36062127